CLINICAL TRIAL: NCT01368055
Title: An Expanded Phase II Study of Hypofractionated Dose Intense Image Guided Proton Radiation Therapy for Low and Intermediate Risk Adenocarcinoma of the Prostate
Brief Title: Hypofractionated Proton Radiation Therapy for Low and Intermediate Risk Prostate Cancer
Acronym: PR07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 1103-PR07; IRB201701768 (Other: University of Florida)
Record Dates: First submitted 2011-06-01; First posted 2011-06-07 (Estimated); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Proton Radiation, Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Risk (Experimental): 70 Gy/CGE
  Interventions: Radiation: 70 Gy/CGE
- Intermediate Risk (Experimental): 72.5 Gy/CGE
  Interventions: Radiation: 72.5 Gy/CGE

INTERVENTIONS:
Radiation: 70 Gy/CGE — Low Risk
  Arms: Low Risk
Radiation: 72.5 Gy/CGE — Intermediate Risk
  Arms: Intermediate Risk

SUMMARY:
The purpose of this trial is to give a shorter course (5 ½-6 weeks) of proton radiation that has as little side effects on normal bladder and rectal tissues as the usual longer course (8 weeks) of proton radiation, without decreasing the chance of killing prostate cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer.
* Gleason score 2-6 or 7.
* PSA ≤ 20 ng/ml.

Exclusion Criteria:

* Previous prostate cancer surgery or pelvic radiation.
* Prior/concurrent systemic chemotherapy for prostate cancer.
* Active inflammatory bowel disease (Crohn's disease, diverticulitis or ulcerative colitis) affecting the rectum.
* History of hip replacement.
* Prior intrapelvic surgery.
* Taking Saw Palmetto or methotrexate and unable or unwilling to discontinue its uses during radiation.
* Receiving continuous and current anticoagulation with Warfarin sodium (Coumadin), Clopidogrel bisulfate (Plavix), dabigatran etexilate mesylate (Pradaxa),enoxaparin sodium (Lovenox), or aspirin/er dipyridamole (Aggrenox).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2025-08 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of treatment-related grade 2 or higher rectal bleeding. | 2 years after completion of radiation therapy

SECONDARY OUTCOMES:
Analyzation of quality of life | After radiation: every 6 months for 3 years, then annually for 20 years
Analysis of treatment-related morbidity | Cumulative incidence up to 20 years after completion of radiation therapy
Analysis of disease control | Cumulative incidence up to 20 years after completion of radiation therapy
  Proportion of patients with disease control after completion of treatment
Analysis of overall survival | Cumulative incidence up to 20 years after completion of radiation therapy
  Proportion of patients alive after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Bryant, MD, MPH, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] American Cancer Society. 2010. Ref Type: Electronic Citation
- [Background] Soloway MS, Pareek K, Sharifi R, Wajsman Z, McLeod D, Wood DP Jr, Puras-Baez A; Lupron Depot Neoadjuvant Prostate Cancer Study Group. Neoadjuvant androgen ablation before radical prostatectomy in cT2bNxMo prostate cancer: 5-year results. J Urol. 2002 Jan;167(1):112-6. PMID 11743286
- [Background] Hull GW, Rabbani F, Abbas F, Wheeler TM, Kattan MW, Scardino PT. Cancer control with radical prostatectomy alone in 1,000 consecutive patients. J Urol. 2002 Feb;167(2 Pt 1):528-34. doi: 10.1016/S0022-5347(01)69079-7. PMID 11792912
- [Background] Kestin LL, Martinez AA, Stromberg JS, Edmundson GK, Gustafson GS, Brabbins DS, Chen PY, Vicini FA. Matched-pair analysis of conformal high-dose-rate brachytherapy boost versus external-beam radiation therapy alone for locally advanced prostate cancer. J Clin Oncol. 2000 Aug;18(15):2869-80. doi: 10.1200/JCO.2000.18.15.2869. PMID 10920135
- [Background] Merrick GS, Butler WM, Wallner KE, Galbreath RW, Allen ZA, Adamovich E. The impact of primary Gleason grade on biochemical outcome following brachytherapy for hormone-naive Gleason score 7 prostate cancer. Cancer J. 2005 May-Jun;11(3):234-40. doi: 10.1097/00130404-200505000-00010. PMID 16053667
- [Background] Demanes DJ, Rodriguez RR, Schour L, Brandt D, Altieri G. High-dose-rate intensity-modulated brachytherapy with external beam radiotherapy for prostate cancer: California endocurietherapy's 10-year results. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1306-16. doi: 10.1016/j.ijrobp.2004.08.014. PMID 15817332
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Common Terminology Criteria for Adverse Events (CTCAE). National Cancer Institute. 12-12-0003. 9-9-0005. Ref Type: Electronic Citation
- [Background] Chism DB, Hanlon AL, Horwitz EM, Feigenberg SJ, Pollack A. A comparison of the single and double factor high-risk models for risk assignment of prostate cancer treated with 3D conformal radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):380-5. doi: 10.1016/j.ijrobp.2003.10.059. PMID 15145151
- [Background] Martinez AA, Demanes DJ, Galalae R, Vargas C, Bertermann H, Rodriguez R, Gustafson G, Altieri G, Gonzalez J. Lack of benefit from a short course of androgen deprivation for unfavorable prostate cancer patients treated with an accelerated hypofractionated regime. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1322-31. doi: 10.1016/j.ijrobp.2004.12.053. PMID 16029788
- [Background] Roach M, Lu J, Pilepich MV, Asbell SO, Mohiuddin M, Terry R, Grignon D. Four prognostic groups predict long-term survival from prostate cancer following radiotherapy alone on Radiation Therapy Oncology Group clinical trials. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):609-15. doi: 10.1016/s0360-3016(00)00578-2. PMID 10837943
- [Background] Ghilezan MJ, Jaffray DA, Siewerdsen JH, Van Herk M, Shetty A, Sharpe MB, Zafar Jafri S, Vicini FA, Matter RC, Brabbins DS, Martinez AA. Prostate gland motion assessed with cine-magnetic resonance imaging (cine-MRI). Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):406-17. doi: 10.1016/j.ijrobp.2003.10.017. PMID 15890582
- [Background] Padhani AR, Khoo VS, Suckling J, Husband JE, Leach MO, Dearnaley DP. Evaluating the effect of rectal distension and rectal movement on prostate gland position using cine MRI. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):525-33. doi: 10.1016/s0360-3016(99)00040-1. PMID 10348281
- [Background] Litzenberg D, Dawson LA, Sandler H, Sanda MG, McShan DL, Ten Haken RK, Lam KL, Brock KK, Balter JM. Daily prostate targeting using implanted radiopaque markers. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):699-703. doi: 10.1016/s0360-3016(01)02654-2. PMID 11849792
- [Background] Litzenberg DW, Balter JM, Hadley SW, Sandler HM, Willoughby TR, Kupelian PA, Levine L. Influence of intrafraction motion on margins for prostate radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):548-53. doi: 10.1016/j.ijrobp.2005.12.033. Epub 2006 Mar 20. PMID 16545919
- [Background] Vargas C, Yan D, Kestin LL, Krauss D, Lockman DM, Brabbins DS, Martinez AA. Phase II dose escalation study of image-guided adaptive radiotherapy for prostate cancer: use of dose-volume constraints to achieve rectal isotoxicity. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):141-9. doi: 10.1016/j.ijrobp.2004.12.017. PMID 16111582
- [Background] Vargas C, Martinez A, Kestin LL, Yan D, Grills I, Brabbins DS, Lockman DM, Liang J, Gustafson GS, Chen PY, Vicini FA, Wong JW. Dose-volume analysis of predictors for chronic rectal toxicity after treatment of prostate cancer with adaptive image-guided radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1297-308. doi: 10.1016/j.ijrobp.2004.12.052. PMID 16029785
- [Background] Dearnaley DP, Hall E, Lawrence D, Huddart RA, Eeles R, Nutting CM, Gadd J, Warrington A, Bidmead M, Horwich A. Phase III pilot study of dose escalation using conformal radiotherapy in prostate cancer: PSA control and side effects. Br J Cancer. 2005 Feb 14;92(3):488-98. doi: 10.1038/sj.bjc.6602301. PMID 15685244
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Sathya JR, Davis IR, Julian JA, Guo Q, Daya D, Dayes IS, Lukka HR, Levine M. Randomized trial comparing iridium implant plus external-beam radiation therapy with external-beam radiation therapy alone in node-negative locally advanced cancer of the prostate. J Clin Oncol. 2005 Feb 20;23(6):1192-9. doi: 10.1200/JCO.2005.06.154. PMID 15718316
- [Background] Shipley WU, Verhey LJ, Munzenrider JE, Suit HD, Urie MM, McManus PL, Young RH, Shipley JW, Zietman AL, Biggs PJ, et al. Advanced prostate cancer: the results of a randomized comparative trial of high dose irradiation boosting with conformal protons compared with conventional dose irradiation using photons alone. Int J Radiat Oncol Biol Phys. 1995 Apr 30;32(1):3-12. doi: 10.1016/0360-3016(95)00063-5. PMID 7721636
- [Background] Vargas, C, Martinez, A, and Boike, T. Long term survival benefit of a prospective dose escalation trial using high dose rate (HDR) brachytherapy boost. Int.J.Radiat.Oncol.Biol.Phys.2005.
- [Background] Vargas C, Martinez A, Galalae R, Demanes J, Harsolia A, Schour L, Nuernberg N, Gonzalez J. High-dose radiation employing external beam radiotherapy and high-dose rate brachytherapy with and without neoadjuvant androgen deprivation for prostate cancer patients with intermediate- and high-risk features. Prostate Cancer Prostatic Dis. 2006;9(3):245-53. doi: 10.1038/sj.pcan.4500882. Epub 2006 Jun 20. PMID 16786040
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Kupelian PA, Reddy CA, Klein EA, Willoughby TR. Short-course intensity-modulated radiotherapy (70 GY at 2.5 GY per fraction) for localized prostate cancer: preliminary results on late toxicity and quality of life. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):988-93. doi: 10.1016/s0360-3016(01)01730-8. PMID 11704322
- [Background] Kupelian PA, Reddy CA, Carlson TP, Altsman KA, Willoughby TR. Preliminary observations on biochemical relapse-free survival rates after short-course intensity-modulated radiotherapy (70 Gy at 2.5 Gy/fraction) for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2002 Jul 15;53(4):904-12. doi: 10.1016/s0360-3016(02)02836-5. PMID 12095556
- [Background] Kupelian PA, Thakkar VV, Khuntia D, Reddy CA, Klein EA, Mahadevan A. Hypofractionated intensity-modulated radiotherapy (70 gy at 2.5 Gy per fraction) for localized prostate cancer: long-term outcomes. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1463-8. doi: 10.1016/j.ijrobp.2005.05.054. Epub 2005 Sep 19. PMID 16169683
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Bush DA, Jabola BR, Levy RP, Grove RI, Preston W, Slater JM. Proton therapy for prostate cancer: the initial Loma Linda University experience. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):348-52. doi: 10.1016/j.ijrobp.2003.10.011. PMID 15145147
- [Background] Ehrenpreis ED, Jani A, Levitsky J, Ahn J, Hong J. A prospective, randomized, double-blind, placebo-controlled trial of retinol palmitate (vitamin A) for symptomatic chronic radiation proctopathy. Dis Colon Rectum. 2005 Jan;48(1):1-8. doi: 10.1007/s10350-004-0821-7. PMID 15690650
- [Background] Denton A, Forbes A, Andreyev J, Maher EJ. Non surgical interventions for late radiation proctitis in patients who have received radical radiotherapy to the pelvis. Cochrane Database Syst Rev. 2002;(1):CD003455. doi: 10.1002/14651858.CD003455. PMID 11869662
- [Background] Cavcic J, Turcic J, Martinac P, Jelincic Z, Zupancic B, Panijan-Pezerovic R, Unusic J. Metronidazole in the treatment of chronic radiation proctitis: clinical trial. Croat Med J. 2000 Sep;41(3):314-8. PMID 10962052
- [Background] Delanian S, Lefaix JL. Current management for late normal tissue injury: radiation-induced fibrosis and necrosis. Semin Radiat Oncol. 2007 Apr;17(2):99-107. doi: 10.1016/j.semradonc.2006.11.006. PMID 17395040
- [Background] Lefaix JL, Delanian S, Vozenin MC, Leplat JJ, Tricaud Y, Martin M. Striking regression of subcutaneous fibrosis induced by high doses of gamma rays using a combination of pentoxifylline and alpha-tocopherol: an experimental study. Int J Radiat Oncol Biol Phys. 1999 Mar 1;43(4):839-47. doi: 10.1016/s0360-3016(98)00419-2. PMID 10098440
- [Background] Delanian S, Porcher R, Balla-Mekias S, Lefaix JL. Randomized, placebo-controlled trial of combined pentoxifylline and tocopherol for regression of superficial radiation-induced fibrosis. J Clin Oncol. 2003 Jul 1;21(13):2545-50. doi: 10.1200/JCO.2003.06.064. PMID 12829674
- [Background] Spry N, Halkett G, Aoun S, Spry J, Yeoh E. Development of a European organization for research and treatment of cancer module to assess the quality of life of patients with proctitis after pelvic radiotherapy for malignancy. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):522-8. doi: 10.1016/j.ijrobp.2007.12.062. Epub 2008 Apr 18. PMID 18374505
- [Background] Freeman DE, King CR. Stereotactic body radiotherapy for low-risk prostate cancer: five-year outcomes. Radiat Oncol. 2011 Jan 10;6:3. doi: 10.1186/1748-717X-6-3. PMID 21219625
- [Background] Vargas C, Fryer A, Mahajan C, Indelicato D, Horne D, Chellini A, McKenzie C, Lawlor P, Henderson R, Li Z, Lin L, Olivier K, Keole S. Dose-volume comparison of proton therapy and intensity-modulated radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Mar 1;70(3):744-51. doi: 10.1016/j.ijrobp.2007.07.2335. Epub 2007 Sep 27. PMID 17904306
- [Background] Michalski JM, Bae K, Roach M, Markoe AM, Sandler HM, Ryu J, Parliament MB, Straube W, Valicenti RK, Cox JD. Long-term toxicity following 3D conformal radiation therapy for prostate cancer from the RTOG 9406 phase I/II dose escalation study. Int J Radiat Oncol Biol Phys. 2010 Jan 1;76(1):14-22. doi: 10.1016/j.ijrobp.2009.01.062. PMID 19577865
- [Background] McGowan, D, Hunt, D, Jones, C, et al. Effect of short-term endocrine therapy prior to and during radiation therapy on overall survival in patients with T1b-T2b adenocarcinoma of the prostate and PSA equal to or less than 20: Initial results of RTOG 94-08 (abstract). American Society of Clinical Oncology (ASCO) 2010 Genitourinary Cancers Symposium. (Abstract available online: http://www.asco.org/ASCOv2/Meetings/Abstracts?&vmview=abst_meeting_categories_view&confID=73, accessed on March 19, 2010).
- [Background] Roach M 3RD, Lu J, Pilepich MV, Asbell SO, Mohiuddin M, Terry R, Grignon D, Lawton C, Shipley W, Cox J. Predicting long-term survival, and the need for hormonal therapy: a meta-analysis of RTOG prostate cancer trials. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):617-27. doi: 10.1016/s0360-3016(00)00577-0. PMID 10837944
- [Background] Arcangeli G, Saracino B, Gomellini S, Petrongari MG, Arcangeli S, Sentinelli S, Marzi S, Landoni V, Fowler J, Strigari L. A prospective phase III randomized trial of hypofractionation versus conventional fractionation in patients with high-risk prostate cancer. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):11-8. doi: 10.1016/j.ijrobp.2009.07.1691. Epub 2010 Jan 4. PMID 20047800
- [Background] Kupelian PA, Willoughby TR, Reddy CA, Klein EA, Mahadevan A. Hypofractionated intensity-modulated radiotherapy (70 Gy at 2.5 Gy per fraction) for localized prostate cancer: Cleveland Clinic experience. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1424-30. doi: 10.1016/j.ijrobp.2007.01.067. Epub 2007 Jun 4. PMID 17544601
- [Background] Mendenhall NP, Li Z, Hoppe BS, Marcus RB Jr, Mendenhall WM, Nichols RC, Morris CG, Williams CR, Costa J, Henderson R. Early outcomes from three prospective trials of image-guided proton therapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):213-21. doi: 10.1016/j.ijrobp.2010.09.024. Epub 2010 Nov 17. PMID 21093164
- [Background] Coote JH, Wylie JP, Cowan RA, Logue JP, Swindell R, Livsey JE. Hypofractionated intensity-modulated radiotherapy for carcinoma of the prostate: analysis of toxicity. Int J Radiat Oncol Biol Phys. 2009 Jul 15;74(4):1121-7. doi: 10.1016/j.ijrobp.2008.09.032. Epub 2009 Jan 7. PMID 19131179
- [Background] Martin JM, Rosewall T, Bayley A, Bristow R, Chung P, Crook J, Gospodarowicz M, McLean M, Menard C, Milosevic M, Warde P, Catton C. Phase II trial of hypofractionated image-guided intensity-modulated radiotherapy for localized prostate adenocarcinoma. Int J Radiat Oncol Biol Phys. 2007 Nov 15;69(4):1084-9. doi: 10.1016/j.ijrobp.2007.04.049. Epub 2007 Jul 2. PMID 17606331
- [Background] Friedland JL, Freeman DE, Masterson-McGary ME, Spellberg DM. Stereotactic body radiotherapy: an emerging treatment approach for localized prostate cancer. Technol Cancer Res Treat. 2009 Oct;8(5):387-92. doi: 10.1177/153303460900800509. PMID 19754215
- [Background] King CR, Brooks JD, Gill H, Pawlicki T, Cotrutz C, Presti JC Jr. Stereotactic body radiotherapy for localized prostate cancer: interim results of a prospective phase II clinical trial. Int J Radiat Oncol Biol Phys. 2009 Mar 15;73(4):1043-8. doi: 10.1016/j.ijrobp.2008.05.059. Epub 2008 Aug 26. PMID 18755555
- [Background] Dearnaley DP, Sydes MR, Graham JD, Aird EG, Bottomley D, Cowan RA, Huddart RA, Jose CC, Matthews JH, Millar J, Moore AR, Morgan RC, Russell JM, Scrase CD, Stephens RJ, Syndikus I, Parmar MK; RT01 collaborators. Escalated-dose versus standard-dose conformal radiotherapy in prostate cancer: first results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2007 Jun;8(6):475-87. doi: 10.1016/S1470-2045(07)70143-2. PMID 17482880
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Peeters ST, Heemsbergen WD, Koper PC, van Putten WL, Slot A, Dielwart MF, Bonfrer JM, Incrocci L, Lebesque JV. Dose-response in radiotherapy for localized prostate cancer: results of the Dutch multicenter randomized phase III trial comparing 68 Gy of radiotherapy with 78 Gy. J Clin Oncol. 2006 May 1;24(13):1990-6. doi: 10.1200/JCO.2005.05.2530. PMID 16648499
- See also: (Contact the University of Florida Proton Therapy Institute) — https://www.floridaproton.org/about-us/contact-us